CLINICAL TRIAL: NCT00781105
Title: An Open-label, Multicenter, Phase IV Study to Evaluate the Efficacy and Safety of Telbivudine 600mg Tablets in Chinese Patients With Chronic Hepatitis B
Brief Title: Efficacy and Safety of Telbivudine 600mg Tablets in Chinese Patients With Chronic Hepatitis B
Acronym: Chinese PAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600ACN03
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; Adult; HBV DNA suppression; Telbivudine
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Telbivudine

INTERVENTIONS:
Drug: Telbivudine — 600 mg/day, oral tablets, once daily, 52 weeks

SUMMARY:
The "Chinese PAC" study (CLDT600ACN03) will evaluate the efficacy and safety of open label telbivudine in 2,200 compensated Chronic Hepatitis B (CHB) adults. The primary objective of the study is the proportion of patients achieving undetectable HBV DNA at week 52.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 16 to 65 year of age
* Documented CHB defined by detectable serum HBsAg and serum HBV DNA level
* Willing and able to comply with the study drug regimen
* Written informed consent before any assessment

Exclusion Criteria:

* Patient has a history of/or clinical signs/symptoms of hepatic decompensation
* Patient has a history of HCC or findings suggestive of possible HCC
* Patient has received treatment of nucleoside or nucleotide drugs whether approved or investigational at any time
* History of hypersensitivity to any of the drugs (telbivudine) or to drugs of similar clinical classes
* Patient has received IFN or other immunomodulatory treatment with 12 months before screening
* Previous treatment history with NRTIs

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2200 (Actual)
Dates: Start 2008-08-01 (Actual); Primary Completion 2010-09-16 (Actual); Study Completion 2010-09-16 (Actual)

PRIMARY OUTCOMES:
HBV DNA PCR negativity rate | at 52 weeks

SECONDARY OUTCOMES:
HBV DNA PCR negativity rate | at week 24
DNA reduction | from baseline to Weeks 12, 24, 36, 52
HBeAg loss rate | at week 52
HBeAg seroconversion rate | at week 52
ALT normalization rate | at weeks 24 and 52
Incidence of AE (SAE,etc), Graded lab abnormalities | at week 52

CONTACTS AND LOCATIONS:
Overall Officials: Jia Jidong, Dr., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Novartis Investigative Site, Beijing, China